CLINICAL TRIAL: NCT00244231
Title: A Placebo-Controlled, Double Blind Study to Evaluate the Efficacy and Safety of Nidadd in the Management of Hyperlipidemia
Brief Title: Efficacy and Safety Study of Nidadd in the Management of Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBL03-NSR
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Hyperlipidemia
Keywords: Niacin; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nidadd

SUMMARY:
To assess the efficacy and safety of Nidadd (extended-release niacin) in patients with hyperlipidemia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, and multicenter study. A total of at least 50 patients will be recruited to achieve 40 evaluable patients required to assess the safety and efficacy of escalating doses of extended-release Nidadd in hyperlipidemic patients.

1. The trial begins with measurement of baseline lipid levels. Fasting blood samples will be collected at screening and each treatment visit (except visit 3) for lipid analysis and safety monitoring. Chemistry laboratory tests and hematological testing are performed periodically. Patient's diet education will be given by dieticians or appropriately trained counselors at visit 1 and 2.
2. Patients who are taking any lipid-modifying drugs will be required to go through a 4-week washout / diet-controlled period prior to randomization (visit 2).
3. Treatment duration is 16 weeks in total: Patients randomized to treatment with Nidadd will receive 500 mg for the first 8 weeks of the medication period. For another 8 weeks, the dose is then increased to 1000 mg and is maintained to the end of the study. The patients in control group will take placebo in a same fashion as that of Nidadd group throughout entire 16 weeks.
4. The primary measure of efficacy is the change from baseline in serum HDL-c level. Secondary measures of efficacy are changes from baseline in serum total cholesterol, LDL-c, and triglycerides.
5. Safety and tolerability will be evaluated from adverse events, number of patients who prematurely discontinue the trial because of adverse events, and laboratory measures.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 20 and 75 years.
2. An at least 4 weeks wash-out / diet-controlled period before study entry is required.
3. HDL cholesterol < 40 mg/dL for male and < 50 mg/dL for female; and triglyceride levels ≧ 200 mg/dL.
4. Being mentally competent and able to understand all study requirements and sign the informed consent form.

Exclusion Criteria:

1. Total cholesterol ≧ 300 mg/dL; triglyceride levels ≧ 1000 mg/dL.
2. Having FPG level greater than 180 mg/dL after a 4-week washout / diet control period.
3. Type-1 diabetes mellitus; or type-2 diabetes mellitus without stable (fixed dose) medication.
4. Pregnant or lactating women or women of childbearing potential whom are not practicing a reliable form of birth control (either with IUD or with stable usage of oral contraceptives).
5. Concomitant steroid therapy.
6. Received any lipid-modifying agents within the four weeks of wash-out / diet-controlled period.
7. With clinically significant cardiac arrhythmias or other serious cardiac abnormalities; received coronary artery bypass graft or percutaneous transluminal coronary angioplasty within 6 months prior to study entry.
8. Malignant tumor (except for squamous/basal cell skin cancer), or chronic terminal disease (e.g. AIDS, liver cirrhosis, etc.) within past 5 years.
9. With any disorders or conditions which, in the opinion of the investigator will preclude successful compliant participation in the study.
10. Nephrotic syndrome or any other renal dysfunction, serum creatinine > 2.0 mg/dl; active hepatic dysfunction, SGPT, SGOT, gGT, or alkaline phosphatase value greater than 2 times the upper limit of normal.
11. With pancreatitis, gallbladder disease, or active peptic ulcer disease within 6 months.
12. Active gouty arthritis.
13. Taken any other investigational drug within one month prior to study entry.
14. With known hypersensitivity to niacin.
15. With a history of alcohol and/or drug abuse.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-10; Study Completion 2005-08

PRIMARY OUTCOMES:
Change from baseline in HDL-c levels

SECONDARY OUTCOMES:
Changes from baseline in serum total cholesterol , LDL-c, and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Der Lin, M.D., Principal Investigator — Chang GungMemorial Hospital; Jawl-Shan Huang, M.D., Principal Investigator — Chang Gung Memorial Hospital; Miaw-jene Liou, M.D., Principal Investigator — Chang Gung Memorial Hospital; Chih-ching Wang, M.D., Principal Investigator — Chang Gung Memorial Hospital; Yi-Jen Hung, M.D., Principal Investigator — Tri-Service General Hospital; Chang-Hsun Hsieh, M.D., Principal Investigator — Tri-Service General Hospital; Chih-Tsueng He, M.D., Principal Investigator — Tri-Service General Hospital; Huey-Herng Sheu, M.D., Principal Investigator — Taichung Veterans General Hospital; Yu-Ling Lin, M.D., Principal Investigator — Taichung Veterans General Hospital; Shih-Yi Lin, M.D., Principal Investigator — Taichung Veterans General Hospital; Yih-Jing Tang, M.D., Principal Investigator — Taichung Veterans General Hospital